CLINICAL TRIAL: NCT01990235
Title: Improving Advance Care Planning by Preparing Diverse Seniors for Decision Making
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13-10847; R01AG045043 (NIH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-21 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Chronic Disease
Keywords: Advance care planning; Aging; Health communication; Health literacy; Medical decision making; primary care; vulnerable population; chronic illness
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PREPARE intervention (Experimental): The PREPARE arm will review the PREPARE website plus the easy-to-read advance directive (AD). Participants will review PREPARE on their own for ≥ 20 minutes with staff present to answer questions. During PREPARE, participants answer preference questions and make an action plan (i.e., commitment to engage in advance care planning). To ensure home access to PREPARE content, participants will be given a website login and PREPARE content in digital video disc (DVD), booklet, and pamphlet format as well as the action plan and AD. One to three days before a primary care visit, the PREPARE arm will receive a reminder to come to their appointment and to bring their action plan.
  Interventions: Behavioral: PREPARE Intervention
- Control (No Intervention): The Control arm will review an easy-to-read AD. Controls will review the AD for ≥ 15 minutes with study staff present to answer questions and will take the AD home to complete if desired. One to three days before a primary care visit, controls will receive a reminder to come to their appointment.

INTERVENTIONS:
Behavioral: PREPARE Intervention — At week 1, 3, 6, and 12 months, interviews (telephone or in person based on preference) by blinded staff will assess engagement in advance care planning(ACP), self-efficacy with ACP, and activation in and satisfaction with decision making. Blinded telephone interviews will also assess surrogate reports of patient engagement in ACP.
  Arms: PREPARE intervention

SUMMARY:
The objective of this proposal is to test whether a multi-media website (www.prepareforyourcare.org) that is focused on preparing older adults for communication and medical decision making can help people engage in advance care planning.

DETAILED DESCRIPTION:
PREPARE is a website (www.prepareforyourcare.org) that teaches patients how to identify what is most important in life, how to communicate their preferences to clinicians and loved ones, and how to make informed decisions. It is written at a 5th grade level and includes voice-overs of text and closed captioning of videos that model advance care planning behaviors. The goal of this proposal is to test the efficacy of PREPARE plus an easy-to-read advance directive, versus an advance directive alone, to improve patient engagement in multiple advance care planning behaviors including discussions with surrogate decision makers and clinicians in addition to advance directive completion. The investigators will also determine whether PREPARE can empower and activate patients within clinical encounters with their clinicians and help to decrease health disparities in advance care planning.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking older adults (≥55 years)
* ≥ 2 chronic illnesses determined by International Classification of Diseases-9 (ICD-9) codes
* ≥ 2 visits with an outpatient primary care clinician at San Francisco General Hospital in the past year
* ≥2 additional outpatient/inpatient visits to San Francisco General Hospital in the past year

Exclusion Criteria:

* deaf, blind, or demented as determined by ICD-9 codes
* too mentally or physically ill to participate as determined by their clinicians
* Moderate or severe cognitive impairment as determined by the Short Portable Mental Status Questionnaire (SPMSQ), and mild cognitive impairment as determined by the SPMSQ plus an abnormal Mini-Cog
* self-reported poor vision and inability to see the words on a newspaper
* lack of a telephone
* traveling or moving out of the area for ≥3 months during the study follow- up period

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2013-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
New advance care planning documentation in the medical record | 15 months after study enrollment
  The primary outcome is documentation of ACP wishes in the medical record. ACP documentation for the purposes of this study includes legal advance directive forms or other documentation of patients wishes for medical care in clinical notes.

SECONDARY OUTCOMES:
Self-reported engagement in advance care planning behaviors | 12 months from baseline
  Secondary outcomes were chosen to measure the full process of ACP. Using validated questionnaires, we will measure ACP behavior change processes, such as knowledge, contemplation, self-efficacy, and readiness, as well as several ACP actions, such as identifying a surrogate decision maker, identifying values and goals for medical care, choosing the level of leeway in surrogate decision making, discussing one's wishes with clinicians and surrogates, and documenting one's wishes in an advance directive.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sudore, MD, Principal Investigator — University of California, San Francisco; Dean Schillinger, MD, Principal Investigator — University of California, San Francisco; Deborah E Barnes, PhD, Principal Investigator — University of California, San Francisco; W. John Boscardin, PhD, Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco General Hospital and Trauma Center, San Francisco, California, United States

REFERENCES:
- [Derived] Gelfman LP, Barnes DE, Goldstein N, Volow AM, Shi Y, Li B, Sudore RL. Quality and Satisfaction With Advance Care Planning Conversations Among English- and Spanish-Speaking Older Adults. J Palliat Med. 2023 Oct;26(10):1380-1385. doi: 10.1089/jpm.2022.0565. Epub 2023 Jun 19. PMID 37335910
- [Derived] Freytag J, Street RL Jr, Barnes DE, Shi Y, Volow AM, Shim JK, Alexander SC, Sudore RL. Empowering Older Adults to Discuss Advance Care Planning During Clinical Visits: The PREPARE Randomized Trial. J Am Geriatr Soc. 2020 Jun;68(6):1210-1217. doi: 10.1111/jgs.16405. Epub 2020 Mar 10. PMID 32157684
- [Derived] Sudore RL, Schillinger D, Katen MT, Shi Y, Boscardin WJ, Osua S, Barnes DE. Engaging Diverse English- and Spanish-Speaking Older Adults in Advance Care Planning: The PREPARE Randomized Clinical Trial. JAMA Intern Med. 2018 Dec 1;178(12):1616-1625. doi: 10.1001/jamainternmed.2018.4657. PMID 30383086
- [Derived] Sudore RL, Barnes DE, Le GM, Ramos R, Osua SJ, Richardson SA, Boscardin J, Schillinger D. Improving advance care planning for English-speaking and Spanish-speaking older adults: study protocol for the PREPARE randomised controlled trial. BMJ Open. 2016 Jul 11;6(7):e011705. doi: 10.1136/bmjopen-2016-011705. PMID 27401363
- See also: PREPARE — http://www.prepareforyourcare.org